CLINICAL TRIAL: NCT06267170
Title: A Multicenter, Real-world Study of Adebrelimab in the Treatment of Extensive Stage
Brief Title: A Multicenter, Real-world Study of Adebrelimab in the Treatment of Extensive Stage Small Cell Lung Cancer
Acronym: SCLC
Status: Not yet recruiting | Type: Observational
Sponsor: Henan Cancer Hospital (Other Government)
Responsible Party: Principal Investigator, Qiming Wang, Chief physician, Henan Cancer Hospital
Other Study IDs: SCLC-RWS-001
Record Dates: First submitted 2024-01-30; First posted 2024-02-20 (Actual); Last update posted 2024-02-20 (Actual); Status verified 2024-02

CONDITIONS: SCLC,Extensive Stage

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Drug: Adebrelimab — Treatment with adbelizumab

SUMMARY:
This study collected data on patients with extensive stage small cell lung cancer treated with Adebrelimab to investigate its safety and efficacy

ELIGIBILITY:
Inclusion Criteria:

1. Sign informed consent and join the study voluntarily;
2. Patients diagnosed with extensive small cell lung cancer;
3. Age ≥18 years old;
4. Have at least one measurable lesion (according to RECIST 1.1);
5. The investigators judged that adebrelimab treatment was acceptable;
6. Contraception: Patients should agree that it must be used during the study period and within 6 months after the study ends Effective contraception;

Exclusion Criteria:

1. Allergic to adebrelimab and its excipients;
2. Patients who have also received other immune drugs or therapies;
3. Patients who are participating in other interventional studies;
4. patients with other malignant tumors;
5. Pregnant or lactating women;
6. The investigator considers that the patient is not suitable to participate in any other conditions of the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with extensive stage small cell lung cancer treated with adebrelimab
Sampling Method: Non-Probability Sample
Enrollment: 288 (Estimated)
Dates: Start 2024-02-25 (Estimated); Primary Completion 2025-02-25 (Estimated); Study Completion 2026-02-25 (Estimated)

PRIMARY OUTCOMES:
Safety (Occurrence of ≥ Grade 3 AE) | End of each cycle (each cycle is 28 days)
  The incidence of grade 3 or higher adverse events

SECONDARY OUTCOMES:
PFS | End of every two cycles (each cycle is 28 days)
  Progression free survival
ORR | End of every two cycles (each cycle is 28 days)
  Objective response rate
OS | End of every two cycles (each cycle is 28 days)
  Overall survival
DCR | End of every two cycles (each cycle is 28 days)
  Disease control rate